CLINICAL TRIAL: NCT03025737
Title: Semmelweis Sport - Complex Cardiovascular Screening of Elite, Recreational, Young and Master Athletes
Brief Title: Semmelweis Sport Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: National Research, Development and Innovation Office (NKFIH) of Hungary (K 120277). (Unknown)
Responsible Party: Principal Investigator, Bela Merkely, Principal Investigator, Semmelweis University Heart and Vascular Center
Other Study IDs: Semmelweis Sport
Record Dates: First submitted 2017-01-12; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Athletes Heart
Keywords: Hypertrophy, Left Ventricular; Ventricular Remodeling
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Samples with DNA, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- athletes: Healthy highly trained elite athletes, recreational athletes, young and master athletes free of known structural myocardial disease
- controls: Healthy volunteers without a history of competitive physical exercise

SUMMARY:
The aim of the present proposal is to investigate the development of distinct morphological, functional, biochemical and molecular aspects of short- and long-term sport-induced changes in the heart, to get a better understanding on the (patho)physiology of athlete's heart. The main goal of our research is to deepen our knowledge on the proper differentiation between beneficial (physiological) and harmful (pathological) consequences of professional sport, thereby effectively preventing potential cardiovascular complications of athletes.

DETAILED DESCRIPTION:
CLINICAL METHODS

1. Sport specific questionnaire, patient history and physical examinations - In our detailed questionnaire, specific information is collected about quantity and quality of training, personal and family history and presence of sport specific and general symptoms.
2. Laboratory biochemical examination - Besides the regular routine laboratory parameters, several specific parameters associated with physical exercise are planned to be measured, such as cardiac biomarkers.
3. 12-lead ECG - Resting standard 12-lead digital ECG will be recorded. Extended analysis will be performed according to the latest recommendations.
4. Holter ECG - 24 hour Holter ECG will be recorded. Extended Holter ECG analysis will be performed.
5. Detailed echocardiography
6. Detailed CMR examination
7. Body composition analysis - With a sophisticated bio-electrical impedance analysis, comprehensive whole body composition and hydration analysis will be performed.
8. Cardiopulmonary exercise testing - Sport specific protocols will be used on both treadmill and bike ergometers.

ELIGIBILITY:
Inclusion Criteria:

* age
* no known cardiovascular disease
* history of sport activity (athletes)
* no history of competitive sport (controls)

Exclusion Criteria:

* History of known relevant cardiac disease (including cardiomyopathies)
* Contraindication to MRI or cardiopulmonary exercise testing

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Elite, recreational, young and master athletes Healthy volunteers without a history of competitive physical exercise
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
The primary analysis will be an investigation regarding the athletic adaptation using CMR | Baseline

SECONDARY OUTCOMES:
The primary analysis will be an investigation regarding the athletic adaptation using cardiopulmonary exercise testing | Baseline
The primary analysis will be an investigation regarding the athletic adaptation using resting ECG | Baseline
The primary analysis will be an investigation regarding the athletic adaptation using 24-Hour Holter ECG | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Heart and Vascular Center, Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No